CLINICAL TRIAL: NCT04675437
Title: Impact of Aerobic Exercise Training on Markers of Frailty in Heart Failure and CABG Patients
Brief Title: Impact of Exercise Training on Frailty in CVD Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Professor, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FR-AT-CVD
Record Dates: First submitted 2020-12-07; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Frailty; Cardiovascular Diseases
Keywords: frailty; older adults; cardiovascular diseases; cardiac rehabilitation
MeSH Terms: conditions — Frailty; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Frail patients (CABG, HF or mini-AVR) (Experimental): 12-weeks cardiac exercise program (3 sessions per week) consisting of aerobic exercises (ergometer, treadmill and arm ergometer).
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise — 12-weeks aerobic exercise program

SUMMARY:
The aim of this research project is to examine the impact of aerobic exercise on markers of frailty in patients (of 65 years or older) suffering from heart failure (HF) or after coronary artery bypass grafting (CABG) or mini aortic valve replacement procedures (mini-AVR).

DETAILED DESCRIPTION:
Frailty is defined as a progressive age-related decline in physiological systems that results in decreased reserves of intrinsic capacity, which confers extreme vulnerability to stressors. Based on previous research, there are indications that frailty is highly prevalent in HF, CABG and mini-AVR patients. As a consequence, these patients (both men and women of 65 years or older) will be included in this research project. The 12-week aerobic exercise program (3 sessions per week) will consist of ergometer, treadmill and arm-ergometer exercises. The intensity will be based on the maximal cardiopulmonary exercise test (CPET) of the patient and will correspond with a heart rate between the first and second ventilatory threshold (with a gradual progression over time).

Secondary, correlations will be examined between markers of the CPET and frailty markers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of at least 65 years of age at the start of the study
* To be admitted to Jessa Hospital Hasselt for cardiac rehabilitation after CABG or mini-AVR surgery or because of HF
* Diagnosed as being frail based on the Phenotype of Fried.

Exclusion Criteria:

* A persistently unstable clinical condition (e.g. angina, advanced conduction disturbances, threatening ventricular arrhythmias or acute HF)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-10-20 (Estimated); Study Completion 2021-10-20 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | At baseline (as part of the identification of frailty)
  To examine whether there was a change in body weight (not due to a diet) in the last year
Gait speed | At baseline (as part of the identification of frailty)
  To examine the gait speed based on the 4.6 metres walking test.
Change in gait speed at 12 weeks | 12 weeks
  To examine the change in gait speed based on the 4.6 metres walking test.
Level of physical activity based on the Katz-scale | At baseline (as part of the identification of frailty)
  To examine the level of physical activity based on the Katz-scale (which measures the level of (in)dependence in activities of daily living) (score of 0-6 in which a higher score indicates a better level of physical activity)
Change in level of physical activity at 12 weeks (0-6) (Higher score = better level of physical activity) | 12 weeks
  To examine the change in level of physical activity based on the Katz-scale (which measures the level of (in)dependence in activities of daily living) (score of 0-6 in which a higher score indicates a better level of physical activity)
Exhaustion based on 2 questions of the Center of Epidemiologic Studies Depression Scale (CES-D) | At baseline (as part of the identification of frailty)
  To examine whether the patients suffer from exhaustion based on two questions of the CES-D (in which a score of 2 or 3 on both questions indicates that the patient suffers from exhaustion)
Change in level of exhaustion at 12 weeks based on 2 questions of the Center of Epidemiologic Studies Depression Scale (CES-D) | 12 weeks
  To examine whether there is a change in the level of experienced exhaustion based on two questions of the CES-D (in which a score of 2 or 3 on both questions indicates that the patient suffers from exhaustion)
Handgrip strength | At baseline (as part of the identification of frailty)
  To examine the handgrip strength measured with the Jamar handheld dynamometer.
Change in handgrip strength at 12 weeks | 12 weeks
  To examine the change in handgrip strength measured with the Jamar handheld dynamometer.

SECONDARY OUTCOMES:
Nutritional status based on the Mini Nutritional Assessement (MNA) | At baseline (as part of the identification of frailty)
  To examine the nutritional status based on the MNA (score of 0-30 in which a higher score indicates a better nutritional status)
Change in nutritional status at 12 weeks based on the Mini Nutritional Assessement (MNA) | 12 weeks
  To examine the change in the nutritional status based on the MNA (score of 0-30 in which a higher score indicates a better nutritional status)
Cognitive status based on the Mini Mental State Examination (MMSE) | At baseline (as part of the identification of frailty)
  To examine the cognitive status based on the MMSE (score of 0-30 in which a higher score indicates a better cognitive status)
Change in cognitive status at 12 weeks based on the Mini Mental State Examination (MMSE) | 12 weeks
  To examine the change in cognitive status based on the MMSE (score of 0-30 in which a higher score indicates a better cognitive status)
Physical status/Comorbidities based on the intake of medications | At baseline (as part of the identification of frailty)
  To examine the physical status based on the number of medications (in which a higher level of medication intake / higher number of medications indicates a more worse physical status)
Change in physical status/Comorbidities at 12 weeks based on the intake of medications | 12 weeks
  To examine the change in physical status based on the intake of medications (in which a higher level of medication intake / higher number of medications indicates a more worse physical status)
Psychological status based on the Geriatric Depression Scale (GDS-15) | At baseline (as part of the identification of frailty)
  To examine the psychological status based on the GDS-15 (score of 0-15 in which a higher score indicates a more depressed state)
Change in psychological status at 12 weeks based on the Geriatric Depression Scale (GDS-15) | 12 weeks
  To examine change in the psychological status based on the GDS-15 (score of 0-15 in which a higher score indicates a more depressed state)
Endurance/Balance/Coordination | At baseline (as part of the identification of frailty)
  To examine the endurance, balance and coordination of the patients based on the Timed up and Go Test
Change in endurance/Balance/Coordination at 12 weeks | 12 weeks
  To examine the change in endurance, balance and coordination of the patients based on the Timed up and Go Test

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hansen, Prof. dr., Principal Investigator — Hasselt University
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No